CLINICAL TRIAL: NCT05892107
Title: The Effect of Using Toy and Cartoon Character Masks on Pain and Anxiety During Peripheral Intravenous Catheterization in Children
Brief Title: Effect of Toy and Mask Use on Pain and Anxiety in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Songül OKŞAR, Clinical Nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SNGL03032022
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Intravenous Catheterization
Keywords: Children; Pain; Cartoon Character Mask; Catheterization; Intravenous Catheterization; Anxiety; Toy
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Toy Group (Experimental): 1. Before the toy is given to the child, the child's pre-procedure pain will be assessed with the Wong-Baker Faces Pain Rating Scale.
  2. 2 minutes before the procedure, the parent will be asked to assess the child's pain with VAS (Visual Analog Scale) and their own anxiety level with State Anxiety Inventory.
  3. Body temperature will be measured before the procedure.
  4. Children will be given a toy 1 minute before the procedure.
  5. The child's pain during the procedure will be assessed by the child using the Wong-Baker Faces Pain Rating Scale.
  6. 2 minutes after the procedure, the mother will re-evaluate the child's pain during the procedure using the Visual Analog Scale (VAS) and anxiety during the procedure using the State Anxiety Scale.
  Interventions: Procedure: Toy Group
- Mask group with cartoon characters (Experimental): 1. The child's pain will be assessed with the Wong-Baker Faces Pain Rating Scale before the procedure.
  2. 2 minutes before the procedure, the parent will be asked to assess the child's pain with VAS (Visual Analog Scale) and their own anxiety level with State Anxiety Inventory.
  3. Body temperature will be measured before the procedure.
  4. 1 minute before the procedure, the nurse will greet the child with a mask.
  5. During the procedure, the child's pain will be assessed by the child using the Wong-Baker Faces Pain Rating Scale.
  6. 2 minutes after the procedure, the mother will reassess the child's pain during the procedure using the Visual Analog Scale (VAS) and anxiety during the procedure using the State Anxiety Scale.
  Interventions: Procedure: Mask group with cartoon characters
- Control Group (Active Comparator): 1. Before the procedure, the child's pain will be assessed with the Wong-Baker Faces Pain Rating Scale.
  2. 2 minutes before the procedure, the parent will be asked to assess the child's pain with VAS (Visual Analog Scale) and their own anxiety level with State Anxiety Inventory.
  3. Body temperature will be measured before the procedure.
  4. 1 minute before the procedure, the nurse will greet the child with a white mask on his/her face.
  5. Children in the control group will be subjected to routine procedures (presence of the mother) during blood collection.
  6. During the procedure, the child's pain will be assessed by the child using the Wong-Baker Faces Pain Rating Scale.
  7. 2 minutes after the procedure, the mother will reassess the child's pain during the procedure using the Visual Analog Scale (VAS) and anxiety during the procedure using the State Anxiety Scale.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Toy Group — After meeting the children in the toy group, the toy will be given to the children to play 1 minute before the procedure. Before nonpharmacological interventions in all groups and 2 minutes before the procedure in the control group, the child's pre-procedural pain will be evaluated by explaining the Wong-Baker Faces Pain Rating Scale to the child.
  Arms: Toy Group
Procedure: Mask group with cartoon characters — The nurse who will open the vascular access with the children in the cartoon character mask group will meet the child 1 minute before the procedure with a cartoon character mask on his/her face.In all groups, the mother will be present with the child during the blood collection procedure. Before nonpharmacological interventions in all groups and 2 minutes before the procedure in the control group, the child's pre-procedural pain will be evaluated by explaining the Wong-Baker Faces Pain Rating Scale to the child.
  Arms: Mask group with cartoon characters
Procedure: Control group — In the control group, the nurse who will open the vascular access will meet the child 1 minute before the procedure with a white mask on her/his face. Children in the control group will be subjected to routine procedures before blood collection.In all groups, the mother will be present with the child during the blood collection procedure. Before nonpharmacological interventions in all groups and 2 minutes before the procedure in the control group, the child's pre-procedural pain will be evaluated by explaining the Wong-Baker Faces Pain Rating Scale to the child.
  Arms: Control Group

SUMMARY:
Invasive painful interventions such as diagnostic and therapeutic procedures, blood sampling, injection and vaccine administration are among the greatest fears of children and lead to undesirable experiences both in children and in parents and healthcare personnel due to children's reactions to pain (İnal &Canbulat 2015;Tuna 2014; Wolyniez et al. 2013). It is important for healthcare personnel to spend additional time to manage the child's pain, anxiety and fear of medical procedures (Longobardi et al. 2019, Chen et al. 2020). The American Academy of Pediatrics and the American Pain Society recommend alleviating or minimizing stress and pain, including practices such as venipuncture (Özel &Çetin 2020). Pharmacologic and nonpharmacologic techniques are applied to reduce the emotional and physical effects of painful intervention (Özel &Çetin 2020).

This study was planned to investigate the effect of the nurse's use of a mask with a cartoon character and the child's playing with a sound and light toy on the child's pain and parental anxiety during peripheral intravenous catheterization.

DETAILED DESCRIPTION:
Invasive painful interventions such as diagnostic and therapeutic procedures, blood sampling, injection and vaccine administration are among the greatest fears of children and lead to undesirable experiences both in children and in parents and healthcare personnel due to children's reactions to pain. Especially anxiety, fear and behavioral problems caused by interventional procedures exacerbate children's pain and may prevent the procedure (İnal &Canbulat 2015;Tuna 2014; Wolyniez et al. 2013). It is important for healthcare personnel to spend additional time to manage the child's pain, anxiety and fear of medical procedures (Longobardi et al. 2019, Chen et al. 2020). The American Academy of Pediatrics and the American Pain Society recommend alleviating or minimizing stress and pain, including practices such as venipuncture (Özel &Çetin 2020).

Pain treatment requires a multidisciplinary team approach. One of the indispensable members of this team is the nurse. One of the care philosophies of pediatric nursing is atraumatic care. In this context, reducing the pain of the child and the physical and emotional effects that pain may cause is one of the most important tasks of the nurse (Çöçelli et al. 2008; Semerci et al. 2020).

Pharmacologic and nonpharmacologic techniques are applied to reduce the emotional and physical effects of painful intervention (Özel &Çetin 2020). Nonpharmacologic pain relief methods are preferred because they are both cost-effective and non-invasive and have no risk of side effects (Mohebbi & Azimzadeh 2014). In recent years, research on the use of nonpharmacologic methods by nurses to relieve pain in painful procedures has increased (İnal &Canbulat 2015). Studies have shown that nonpharmacologic methods can be effective alone, especially in pain related to invasive interventions, and when used in combination with pharmacologic methods, they increase the effectiveness of drugs (Uğurlu 2017).

Researchers have reported that the use of distraction technique during painful procedures resulted in less pain reported by children (Dumoulin et al. 2019). In the preschool age group, various distraction activities such as playing with distraction cards, squeezing soft balls, blowing balloons, blowing soap bubbles, playing with dough or Buzzy, guided imagery, and listening to music are utilized ( Chen et al. 2020; Krauss et al. 2016).

In a study in which distraction cards were used during blood sampling, it was found that the use of these cards was effective in relieving pain in children (İnal &Kelleci 2012). In another study conducted to determine the effect of watching cartoons on pain scores and crying duration in children aged 3-6 years during intravenous access, it was found that watching cartoons was a non-pharmacologic pain relief method that decreases pain perception by distracting the child (Akgül et al. 2018).

In a study conducted with children aged 4-6 years, it was found that squeezing a soft ball as a distraction technique could decrease the pain of children during intravenous catheter placement (Sadeghi et al. 2013). In a study conducted to determine the effects of watching animation during blood sampling on pain response in preschool children, statistically significant differences were found in pain, blood cortisol and blood glucose levels in the intervention group (Yoo et al. 2011).

Various masks are used to protect against viruses and bacteria or to avoid infecting people around them. Experts argue that wearing a mask is one of the most effective methods to protect against the coronavirus outbreak during the pandemic process we are in (Ünal &Gökçen 2020). Wearing a mask that will attract the attention and attention of children by healthcare professionals working in pediatric clinics and intervening in children will not frighten the child and may also reduce the perception of procedural pain. It is also thought to be a non-invasive and cost-effective non-pharmacologic intervention to reduce pain.

This study was planned to investigate the effect of the nurse's use of a mask with a cartoon character and the child's playing with a sound and light toy on the child's pain and parental anxiety during peripheral intravenous catheterization.

ELIGIBILITY:
Inclusion Criteria:

* The parent's verbal and written acceptance of the informed consent form,
* The child has not been given any medication with analgesic effect in the last 6 hours,
* Opening the vascular access on the first attempt,
* Body temperature between 36.5-37.2⁰C,
* The child does not have a chronic disease that requires frequent invasive procedures,
* The child does not have a disease that can cause chronic pain,
* The child does not have a mental or neurological disability that would affect participation in the research

Exclusion Criteria:

* Failure of the parent to verbally and in writing accept the informed consent form for participation in the study,
* The child has taken a drug with analgesic, antipyretic, anti-inflammatory effect in the last 6 hours,
* Failure to open the vascular access on the first attempt,
* The child's body temperature is above 37.2⁰C,
* Have a chronic disease that requires frequent invasive procedures,
* The child has a disease that can cause chronic pain,
* The child has an intellectual or neurological disability.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in children's pain level | 2 minutes before the procedure and 2 minutes after the procedure
  The pain level of the children will be evaluated with the Wong Baker Pain Scale.

SECONDARY OUTCOMES:
Parental anxiety score | 2 minutes before the procedure and 2 minutes after the procedure
  The mother's level of anxiety will be scored using the State Anxiety scale.

CONTACTS AND LOCATIONS:
Overall Officials: Birsen MUTLU, Ph.d, Principal Investigator — Istanbul University - Cerrahpasa; Songül OKŞAR, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Songül Okşar, Istanbul, Şişli, Turkey (Türkiye)

REFERENCES:
- [Background] Akgul EA, Karahan Y, Basoglu F, Ogul A, Oztornaci BO, Yetim P, Sari HY. Effects of watching cartoons on pain scores in children undergoing venepuncture. Nurs Child Young People. 2018 Dec 13. doi: 10.7748/ncyp.2018.e913. Online ahead of print. PMID 31468905
- [Background] Chen YJ, Cheng SF, Lee PC, Lai CH, Hou IC, Chen CW. Distraction using virtual reality for children during intravenous injections in an emergency department: A randomised trial. J Clin Nurs. 2020 Feb;29(3-4):503-510. doi: 10.1111/jocn.15088. Epub 2019 Dec 4. PMID 31715039
- [Background] Çöçelli, L. P., Bacaksız, B. D., & Ovayolu, N. (2008). The role of the nurse in pain treatment. Gaziantep Medical Journal, 14(2), 53-58.
- [Background] Dumoulin S, Bouchard S, Ellis J, Lavoie KL, Vezina MP, Charbonneau P, Tardif J, Hajjar A. A Randomized Controlled Trial on the Use of Virtual Reality for Needle-Related Procedures in Children and Adolescents in the Emergency Department. Games Health J. 2019 Aug;8(4):285-293. doi: 10.1089/g4h.2018.0111. Epub 2019 May 24. PMID 31135178
- [Background] Inal, S., Canbulat, N. (2015). The use of distraction methods in procedural pain management in children. Journal of Health Sciences and Professions, 2(3), 372-378.
- [Background] Inal S, Kelleci M. Distracting children during blood draw: looking through distraction cards is effective in pain relief of children during blood draw. Int J Nurs Pract. 2012 Apr;18(2):210-9. doi: 10.1111/j.1440-172X.2012.02016.x. PMID 22435986
- [Background] Krauss BS, Calligaris L, Green SM, Barbi E. Current concepts in management of pain in children in the emergency department. Lancet. 2016 Jan 2;387(10013):83-92. doi: 10.1016/S0140-6736(14)61686-X. Epub 2015 Jun 18. PMID 26095580
- [Background] Longobardi C, Prino LE, Fabris MA, Settanni M. Soap bubbles as a distraction technique in the management of pain, anxiety, and fear in children at the paediatric emergency room: A pilot study. Child Care Health Dev. 2019 Mar;45(2):300-305. doi: 10.1111/cch.12633. Epub 2018 Dec 12. PMID 30466144
- [Background] Mohebbi, P., & Azimzadeh, R. (2014). Barrier of implementing non-pharmacological pain management in children and presented intereventions by nurses. Journal of Holistic Nursing and Midwifery, 24(2), 40-48.
- [Background] Ozel A, Cetin H. [Effects of vibrating tourniquet application on the pain felt for blood drawing in pediatric patients]. Agri. 2020 Jan;32(1):25-30. doi: 10.14744/agri.2019.04900. Turkish. PMID 32030695
- [Background] Semerci R, Kocaaslan EN, Akgun Kostak M, Akin N. [Reduction of pain during intravenous cannulation in children: Buzzy application]. Agri. 2020 Nov;32(4):177-185. doi: 10.14744/agri.2020.02223. Turkish. PMID 33398861
- [Background] Sadeghi T, Mohammadi N, Shamshiri M, Bagherzadeh R, Hossinkhani N. Effect of distraction on children's pain during intravenous catheter insertion. J Spec Pediatr Nurs. 2013 Apr;18(2):109-14. doi: 10.1111/jspn.12018. Epub 2013 Mar 5. PMID 23560582
- [Background] Tuna, P. T. (2014). The effect of practices to prepare for the procedure before peripheral cannula application on pain and anxiety in children (Master's thesis, ESOGÜ, Graduate School of Health Sciences).
- [Background] Wolyniez I, Rimon A, Scolnik D, Gruber A, Tavor O, Haviv E, Glatstein M. The effect of a medical clown on pain during intravenous access in the pediatric emergency department: a randomized prospective pilot study. Clin Pediatr (Phila). 2013 Dec;52(12):1168-72. doi: 10.1177/0009922813502257. Epub 2013 Sep 11. PMID 24028842
- [Background] Yoo H, Kim S, Hur HK, Kim HS. The effects of an animation distraction intervention on pain response of preschool children during venipuncture. Appl Nurs Res. 2011 May;24(2):94-100. doi: 10.1016/j.apnr.2009.03.005. Epub 2009 Jul 15. PMID 20974061
- [Background] Ugurlu, E. S. (2017). Nonpharmacologic pain relief methods in interventional procedures in children. Acıbadem University Journal of Health Sciences, 8(4), 198-201.
- [Background] Ünal, Z., & Gökçen, Ö. (2020). Research on Surgical Masks and Mask Use in Children. Turkish Journal of Fashion Design and Management, 3(1), 11-24.